CLINICAL TRIAL: NCT03001141
Title: Study Protocol/ Registry of MultiPoint™ Pacing in Brazil
Status: Terminated | Type: Observational
Why Stopped: Ethic Comitte (CONEP) determinated the prematurely terminated.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: U1111-1190-5280
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Heart Failure, Unspecified
Keywords: MultiPoint Pacing; Heart Failure; Cardiac Resynchronization Therapy; Quadripolar pacing
MeSH Terms: conditions — Heart Failure | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group - observational
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Device: MultiPoint Pacing will be enabled in enrolled patients at the discretion of the physician.

SUMMARY:
This is a prospective, multicenter, non-randomized registry/observational study. The study will enroll up to 200 patients with successful St. Jude Medical (SJM) Cardiac Resynchronization Therapy (CRT) MP device implant from up to 10 centers.

DETAILED DESCRIPTION:
Any patient receiving a market-approved SJM Quadra Assura MP (CRT-D) or newer model quadripolar device with MPP capability and who meets the inclusion criteria and none of the exclusion criteria is eligible for enrollment in the study.

Patients will be followed for 12 months after implant. Data will be collected after device implant (up to 30 days after successful implant), at 3, 6 and 12 months post-implant and during unscheduled visits.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing and able to sign Informed Consent Form
* Any patient receiving a market-approved SJM Quadra Assura MP (CRT-D) or newer model quadripolar device with MPP capability

Exclusion Criteria:

* Is likely to undergo a heart transplantation within 12 months
* Is less than 18 years old
* Is pregnant or is planning to get pregnant during the study
* Is currently taking part in a Clinical Trial with an active treatment group
* Life expectancy is under 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient receiving a market-approved SJM Quadra Assura MP (CRT-D) or newer model quadripolar device with MPP capability and who meets the inclusion criteria and none of the exclusion criteria is eligible for enrollment in the study.
  Patients will be followed for 12 months after implant. Data will be collected after device implant (up to 30 days after successful implant), at 3, 6 and 12 months post-implant and during unscheduled visits.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Cardiac resynchronization therapy response rate measured by Clinical Composite Score | 12 months
  Evaluated on regular medical visits and registered in the CRF

SECONDARY OUTCOMES:
Quality of Life changes, measured by MLWHF questionnaire | 12 months
  Evaluated on regular medical visits and registered in the CRF
Quality of Life changes, measured by EQ-5D questionnaire | 12 months
  Evaluated on regular medical visits and registered in the CRF
Change in left ventricular ejection fraction | 12 months
  Evaluated on regular medical visits and registered in the CRF
Change in left ventricular end systolic volume | 12 months
  Evaluated on regular medical visits and registered in the CRF
Programming strategy used (vector and intervals), obtained from the Device Session records | 12 months
  Evaluated on regular medical visits and registered in the CRF
Heart failure hospitalization rate | 12 months
  Evaluated on regular medical visits and registered in the CRF
All-cause mortality | 12 months
  Evaluated on regular medical visits and registered in the CRF

CONTACTS AND LOCATIONS:
Overall Officials: Marco Aurelio Santos, Study Director — Abbott Medical Devices
Locations (4):
- Brazil (4):
  - Clinica Dom Rodrigo, João Pessoa, Paraíba
  - BP, São Paulo, São Paulo
  - Instituto de Arritmias Cardíacas, São Paulo, São Paulo
  - SEMAP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided